CLINICAL TRIAL: NCT00124124
Title: A Randomized, Controlled Trial of Melanoma Treatment: Comparison of Dendritic Cells Versus Montanide as Adjuvants to Stimulate Anti-tumor Immunity
Brief Title: Comparison of Dendritic Cells Versus Montanide as Adjuvants in a Melanoma Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Nina Bhardwaj (Individual)
Collaborators: Cancer Research Institute, New York City (Other)
Responsible Party: Sponsor-Investigator, Dr. Nina Bhardwaj, Director, Tumor Vaccine Program, Bhardwaj, Nina, M.D.
Organization: Bhardwaj, Nina, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYU 02-10; NCT00045383 (obsolete NCT alias)
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — keyhole-limpet hemocyanin; Peptides; Monatide (IMS 3015)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): KLH and peptide pulsed DCs
  Interventions: Drug: KLH; Peptides; Dendritic Cells
- 2 (Experimental): KLH, peptides plus Montanide
  Interventions: Drug: KLH, peptides plus Montanide

INTERVENTIONS:
Drug: KLH; Peptides; Dendritic Cells — Upon entry into the study, patients randomized to the dendritic cell arm will undergo a complete baseline evaluation and leukapheresis 0.5 to 3 x 106 DCs per peptide antigen (total not to exceed 18 x 106 cells) will be administered intradermally as per injection SOP. They will receive up to 3 booster DC injections (total not to exceed 18 x 10 6 cells per injection) at monthly intervals for a total of 4 injections. The booster injections will not contain KLH, as our volunteer studies have shown that priming occurs following a single injection of DCs
  Arms: 1
Drug: KLH, peptides plus Montanide — Patients randomized to the Montanide arm will also undergo complete baseline evaluation but not leukapheresis. The peptides will be mixed with the adjuvant, Montanide, and administered subcutaneously at a dose of 100 microgram of each peptide +100 microgram KLH mixed with an equal volume of Montanide. They will receive up to 3 booster injections at monthly intervals for a total of 4 injections. The booster injections will not contain KLH.
  Arms: 2

SUMMARY:
In this study, a melanoma vaccine (5 melanoma peptides) is given with either Montanide or dendritic cells as adjuvants. This randomized trial will establish the safety of both vaccines and compare the 2 vaccine adjuvants in their efficacy to induce immune responses.

DETAILED DESCRIPTION:
In this study, we will examine whether DCs pulsed with candidate melanoma-specific peptides and KLH can boost CTL responses to melanoma antigens in melanoma patients who are clinically free of disease but at high risk for recurrence. This vaccine will be compared to direct injection of the same peptides with KLH and Montanide as adjuvant.

ELIGIBILITY:
Inclusion Criteria:

* Resected stage IIB, IIC, or stage III melanoma.
* Fully recovered from surgery
* Human leukocyte antigen (HLA) A*0201 positive.
* Age >18 years.
* Karnofsky performance status: >80% and normal labs.

Exclusion Criteria:

* Prior chemotherapy.
* Known chronic infection with HIV, hepatitis B or C.
* Patients with known autoimmune disease [e.g. systemic lupus erythematosus (SLE), rheumatoid arthritis (RA)]. Patients with vitiligo are not excluded.
* Pregnant women.
* Patients with known allergy to gentamicin, tobramycin, streptomycin and amikacin (risk of cross-reaction between aminoglycosides).
* Patients who have known retinal or choroidal eye disease.
* Patients previously treated with one of the peptides used in this trial, melanoma protein vaccine, melanoma whole cell vaccines, or with Montanide are not eligible.
* Allergy to shellfish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-07; Primary Completion 2008-07 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Immunology | Examine whether DCs pulsed with candidate melanoma-specific peptides and KLH can boost CTL responses to melanoma antigens

SECONDARY OUTCOMES:
Safety | Post drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Adams, MD, Study Director — NYU Langone Health; Nina Bhardwaj, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Clinical Cancer Center, New York, New York, United States